CLINICAL TRIAL: NCT01091428
Title: Randomized Phase 2 Study of MLN8237, an Aurora A Kinase Inhibitor, Plus Weekly Paclitaxel or Weekly Paclitaxel Alone in Patients With Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer, Preceded by a Phase 1 Portion in Patients With Ovarian or Breast Cancer
Brief Title: Alisertib (MLN8237) in Participants With Ovarian, Fallopian Tube or Peritoneal Cancer Preceded by Phase 1 Study of MLN8237 Plus Paclitaxel Treatment of Ovary or Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C14008; 2009-011428-79 (EudraCT Number); U1111-1191-6584 (Registry Identifier: WHO)
Record Dates: First submitted 2010-03-17; First posted 2010-03-24 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Ovarian Carcinoma; Fallopian Tube Cancer; Peritoneal Cancer; Breast Carcinoma
Keywords: RECIST: Response Evaluation Criteria in Solid Tumors; OC: Ovarian Cancer; GCIG: Gynecologic Cancer Intergroup; Breast carcinoma (Phase 1); Drug therapy
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Breast Neoplasms | interventions — MLN 8237; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Alisertib (Phase 1 - Ovarian cancer) (Experimental): Participants with ovarian cancer received alisertib (MLN8237) 10, 20, 30 or 40 mg, orally, twice daily (BID) on Days 1-3, 8-10 and 15-17, combined with weekly paclitaxel 60 or 80 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 1 (Up to 37 cycles).
  Interventions: Drug: Alisertib; Drug: Paclitaxel
- Alisertib (Phase 1 - Breast cancer) (Experimental): Participants with breast cancer received alisertib (MLN8237) 10, 20, 30 or 40 mg, orally, twice daily (BID) on Days 1-3, 8-10 and 15-17, combined with weekly paclitaxel 60 or 80 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 1 (Up to 37 cycles).
  Interventions: Drug: Alisertib; Drug: Paclitaxel
- Alisertib 40 mg BID+Paclitaxel 60 mg/m^2 (Phase 2) (Experimental): Alisertib 40 mg, orally, BID on Days 1-3, 8-10 and 15-17, combined with weekly paclitaxel 60 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 2 (Up to 28 cycles).
  Interventions: Drug: Alisertib; Drug: Paclitaxel
- Paclitaxel 80 mg/m^2 (Phase 2) (Experimental): Paclitaxel 80 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 2 (Up to 28 cycles).
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Alisertib — Alisertib tablets
  Other Names: MLN8237
  Arms: Alisertib (Phase 1 - Breast cancer); Alisertib (Phase 1 - Ovarian cancer); Alisertib 40 mg BID+Paclitaxel 60 mg/m^2 (Phase 2)
Drug: Paclitaxel — Paclitaxel intravenous infusion

SUMMARY:
This is an open-label, multicenter study with a nonrandomized Phase 1 portion and an open-label, randomized, Phase 2 portion evaluating MLN8237 in combination with weekly paclitaxel in adult female participants with advanced breast cancer (Phase 1 portion only) and recurrent ovarian cancer (both Phase 1 and Phase 2 portions).

DETAILED DESCRIPTION:
The drug tested in this study was called alisertib. Alisertib was tested to treat people who have ovarian and breast cancer. This study looked at safety, any anti-tumor effect, and it also determined a recommended dose of alisertib plus paclitaxel to take into further studies. Pharmacokinetic blood samples were studied to characterize any effects on the concentration of each of the drugs when administered together.

The study enrolled 191 patients. Participants with Breast Cancer and Ovarian Cancer received one of the following escalating doses of alisertib in combination with paclitaxel in the Phase 1 lead-in portion of the study:

* Alisertib 10 mg BID + Paclitaxel 80 mg/m^2
* Alisertib 20 mg BID + Paclitaxel 80 mg/m^2
* Alisertib 20 mg BID + Paclitaxel 60 mg/m^2
* Alisertib 30 mg BID + Paclitaxel 60 mg/m^2
* Alisertib 40 mg BID + Paclitaxel 60 mg/m^2
* Alisertib 50 mg BID + Paclitaxel 60 mg/m^2

Once the maximum tolerated dose (MTD)/ recommended phase 2 dose (RP2D) was determined, participants were randomized to receive the following treatments in the Phase 2 portion of the study:

* Alisertib 40 mg BID + Paclitaxel 60 mg/m^2
* Paclitaxel 80 mg/m^2

This multi-center trial was conducted in the United States, Poland and France. The overall time to participate in this study was approximately 5 years. Participants made multiple visits to the clinic, and who did not experience disease progression (PD) were followed off-treatment once every 8 weeks until the occurrence of 110 progression-free survival (PFS) events.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following inclusion criteria to be enrolled in the study:

* Female participants 18 years or older
* Previously treated, metastatic or locally recurrent malignancy with 1 of the following diagnoses, which has been confirmed histologically or cytologically: adenocarcinoma of the breast (Phase 1 only), recurrent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma (Phase 1 and 2)
* In the Phase 1 portion of the study, participants with breast cancer must have received treatment with at least 1 but no more than 4 prior chemotherapy regimens not including regimens received in the neoadjuvant and/or adjuvant setting
* Participants with breast cancer must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* No antineoplastic therapy or radiotherapy within 3 weeks before enrollment (2 weeks for regimens with recovery expected within 7 to 14 days) and recovered from toxicities of prior therapy (except alopecia); the participant must have recovered from all treatment-related toxicities and must have evidence of progressive disease (PD) or persistent disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate bone marrow, liver and renal function
* Postmenopausal at least 1 year, OR Surgically sterile, OR If childbearing potential, agree to 2 effective methods of nonhormonal contraception, or agree to completely abstain from heterosexual intercourse
* Able to provide written informed consent
* Willing to comply with scheduled visits, treatment plan, laboratory tests and other trial procedures
* Suitable venous access

Specific Inclusion Criteria for participants with Recurrent Ovarian, Fallopian Tube or Peritoneal Cancer:

* Prior treatments must have included a platinum and a taxane; the most recent treatment need not be a platinum-containing or taxane-containing regimen
* Disease must have recurred ≤ 12 months after discontinuation of platinum therapy
* Participants who previously received weekly taxane are potentially eligible, provided that they did not progress during therapy or within 3 months of completing therapy
* Participants with platinum-refractory disease, as defined by progression during primary or subsequent platinum-based therapy or persistent radiographic disease after primary or subsequent platinum-based therapy, will be included
* Participants must have measurable disease in target lesions or assessable disease (defined by cancer antigen-125 - CA-125 per protocol), and disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or modified Gynecologic Cancer Intergroup (GCIG) CA-125 criteria

Exclusion Criteria:

Participants meeting any of the following exclusion criteria are not to be enrolled in the study:

* Prior treatment with an Aurora A-targeted agent (including MLN8237)
* Treatment with clinically significant enzyme inducers within 14 days prior to the first dose of MLN8237 and during the study
* Treatment with more than 4 cytotoxic chemotherapy regimens in the metastatic setting; prior therapy cannot include more than 2 prior taxane-containing regimen. Current use of tamoxifen, thalidomide, or any agent used as maintenance or consolidation therapy for OC.
* Known hypersensitivity to Cremophor® EL, paclitaxel or its components
* Prior history of ≥ Grade 2 neurotoxicity or any toxicity requiring discontinuation from taxane chemotherapy that is not resolved to ≤ Grade 1
* Comorbid or unresolved toxicity that would preclude administration of weekly paclitaxel
* Primary central nervous system malignancy or carcinomatous meningitis
* Symptomatic brain metastasis
* Inability to swallow oral medications or maintain a fast
* History of hemorrhagic or thrombotic cerebrovascular event in past 12 months
* Surgery within 3 weeks before study enrollment and not fully recovered
* Diagnosis or treatment of another malignancy within 2 years preceding first dose of MLN8237 and have any evidence of residual disease except nonmelanoma skin cancer or in situ malignancy completely resected
* Pregnant or lactating
* Serious illness that could interfere with protocol completion
* Investigational treatment 21 days prior to first dose of MLN8237
* Prior allogeneic bone marrow or organ transplantation
* Infection requiring systemic antibiotic therapy within 14 days prior to first dose of MLN8237
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* Radiotherapy to > 25% bone marrow or whole pelvic radiotherapy
* Requirement for constant administration of proton pump inhibitor, H2 antagonist, or pancreatic enzymes. Intermittent uses of antacids of H2 antagonists are allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2010-04-16 (Actual); Primary Completion 2014-08-12 (Actual); Study Completion 2017-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - The Bronx, New York
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Seattle, Washington

REFERENCES:
- [Derived] Falchook G, Coleman RL, Roszak A, Behbakht K, Matulonis U, Ray-Coquard I, Sawrycki P, Duska LR, Tew W, Ghamande S, Lesoin A, Schwartz PE, Buscema J, Fabbro M, Lortholary A, Goff B, Kurzrock R, Martin LP, Gray HJ, Fu S, Sheldon-Waniga E, Lin HM, Venkatakrishnan K, Zhou X, Leonard EJ, Schilder RJ. Alisertib in Combination With Weekly Paclitaxel in Patients With Advanced Breast Cancer or Recurrent Ovarian Cancer: A Randomized Clinical Trial. JAMA Oncol. 2019 Jan 1;5(1):e183773. doi: 10.1001/jamaoncol.2018.3773. Epub 2019 Jan 10. PMID 30347019

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 33 investigative sites in France, Poland and the United States from 16 April 2010 to 19 July 2017. Data cutoff for the primary analysis was 12 August 2014.
Pre-assignment Details: Participants with a diagnosis of ovarian cancer or breast cancer were enrolled equally in a dose escalation study to determine the recommended Phase 2 dose. In Phase 2 participants were randomized equally to receive alisertib 40 mg BID + paclitaxel 60 mg/m^2 or single agent paclitaxel 80 mg/m^2.
Groups:
- Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 (Phase 2): Alisertib 40 mg, orally, BID on Days 1-3, 8-10 and 15-17, combined with weekly paclitaxel 60 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 2 (Up to 28 cycles).
Period: Phase 1
Arm/Group | Alisertib (Phase 1 - Ovarian Cancer) | Alisertib (Phase 1 - Breast Cancer) | Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 (Phase 2) | Paclitaxel 80 mg/m^2 (Phase 2)
Started | 38 | 11 | 0 | 0
Completed | 0 (Completed = participants who completed the treatment.) | 0 | 0 | 0
Not Completed | 38 | 11 | 0 | 0
Not completed — Progressive Disease | 24 | 8 | 0 | 0
Not completed — Symptomatic Deterioration | 3 | 2 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0 | 0
Not completed — Reason not specified | 0 | 1 | 0 | 0
Not completed — Single-Patient IND | 2 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Alisertib (Phase 1 - Ovarian Cancer) | Alisertib (Phase 1 - Breast Cancer) | Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 (Phase 2) | Paclitaxel 80 mg/m^2 (Phase 2)
Started | 0 | 0 | 73 | 69
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 73 | 69
Not completed — Progressive Disease | 0 | 0 | 44 | 46
Not completed — Symptomatic Deterioration | 0 | 0 | 1 | 6
Not completed — Adverse Event | 0 | 0 | 12 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 9 | 8
Not completed — Unsatisfactory Therapeutic Response | 0 | 0 | 1 | 1
Not completed — Reason not specified | 0 | 0 | 4 | 3
Not completed — Physician Decision | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alisertib (Phase 1 - Ovarian Cancer) | Alisertib (Phase 1 - Breast Cancer) | Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 (Phase 2) | Paclitaxel 80 mg/m^2 (Phase 2) | Total
Number analyzed (Participants) | 38 | 11 | 73 | 69 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (10.29) | 58.6 (10.06) | 61.0 (11.60) | 60.8 (8.41) | 59.8 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 11 | 73 | 69 | 191
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 4 | 0 | 1 | 4 | 9
  Not Hispanic or Latino | 34 | 10 | 64 | 62 | 170
  Not Reported | 0 | 1 | 7 | 3 | 11
  Missing | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 34 | 11 | 66 | 55 | 166
  Black or African American | 3 | 0 | 2 | 6 | 11
  Asian | 1 | 0 | 1 | 2 | 4
  American Indian or Alaskan Native | 0 | 0 | 0 | 2 | 2
  Other | 0 | 0 | 1 | 1 | 2
  Not Reported | 0 | 0 | 2 | 3 | 5
  Missing | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 38 | 11 | 48 | 45 | 142
  Poland | 0 | 0 | 10 | 8 | 18
  France | 0 | 0 | 15 | 16 | 31
Height [Mean (Standard Deviation); unit: cm] — Population: Height data was only available for 72 participants in the Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 arm in Phase 2.
  cm
    number analyzed (Participants) | 38 | 11 | 72 | 69 | 190
    (all) | 164.2 (6.41) | 164.5 (6.38) | 162.4 (7.02) | 161.9 (7.30) | 162.7 (6.99)
Weight [Mean (Standard Deviation); unit: kg] | 75.86 (16.41) | 76.29 (7.29) | 70.42 (14.78) | 72.50 (18.71) | 72.59 (16.37)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Body Surface Area (m^2) = square root [height (cm) x weight (kg) / 3600]. Population: Body Surface Area was only calculated for 72 participants in the Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 arm in Phase 2.
  m^2
    number analyzed (Participants) | 38 | 11 | 72 | 69 | 190
    (all) | 1.850 (0.21) | 1.865 (0.10) | 1.776 (0.20) | 1.794 (0.24) | 1.802 (0.21)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) for Alisertib in Combination With Paclitaxel
Description: The MTD is defined as the dose range at which ≤ 1 of 6 evaluable participants experience dose limiting toxicities (DLT). DLT was evaluated according to National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.02 and was defined as any of the following events: 1. Grade 4 neutropenia and thrombocytopenia lasting ≥7 consecutive days; 2. Grade 4 neutropenia with fever and/or infection; 3. Platelet count <10,000/mm^3; 4. Grade 3 thrombocytopenia with bleeding; 5. Any other ≥Grade 3 nonhematologic toxicity, with following exceptions: ≥Grade 3 nausea/emesis, ≥Grade 3 diarrhoea, Grade 3 fatigue, Grade 3 nonhematological toxicity that could be controlled to ≤Grade 2 with appropriate treatment; 6. Other alisertib-related nonhematologic toxicities ≥Grade 2 that, in opinion of investigator, required a dose reduction or discontinuation of therapy with alisertib.
Time Frame: Cycle 1 (Up to 28 days)
Population: DLT-Evaluable Population was defined as all participants in the phase 1 who either experienced DLT during Cycle 1 or completed treatment with at least 15 of the planned 18 doses of alisertib and 2 of the planned 3 doses of paclitaxel in Cycle 1 and had sufficient follow-up data.
Measure: Number; unit: mg
Groups:
- Alisertib + Paclitaxel (Phase 1): Participants with ovarian cancer received alisertib (MLN8237) 10, 20, 30 or 40 mg, orally, twice daily (BID) on Days 1-3, 8-10 and 15-17, combined with weekly paclitaxel 60 or 80 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 1 (Up to 37 cycles).
Arm/Group | Alisertib + Paclitaxel (Phase 1)
Number analyzed (Participants) | 49
mg | 40

2. Primary Outcome: Phase 1: MTD and RP2D for Paclitaxel in Combination With Alisertib
Description: The RP2D is the maximum tolerated dose (MTD) or less. The MTD is defined as the dose range at which ≤ 1 of 6 evaluable participants experience dose limiting toxicities (DLT) within the first 28 days of treatment (end of cycle 1).
Time Frame: Cycle 1 (Up to 28 days)
Population: as for outcome 1
Measure: Number; unit: mg/m^2
Groups:
- Alisertib + Paclitaxel: Paclitaxel 60 or 80 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 1.
Arm/Group | Alisertib + Paclitaxel
Number analyzed (Participants) | 49
mg/m^2 | 60

3. Primary Outcome: Phase 1: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A Serious Adverse Event (SAE) A serious is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: First dose to 30 days past last dose (Up to 36 Months)
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Alisertib (Phase 1 - Ovarian Cancer) | Alisertib (Phase 1 - Breast Cancer)
Number analyzed (Participants) | 38 | 11
participants
  AEs | 38 | 11
  SAEs | 13 | 2

4. Primary Outcome: Phase 1: Number of Participants With Clinically Significant Laboratory Values
Description: Abnormal clinical laboratory values (serum chemistry, hematology and urinalysis) were reported as AEs if they were considered by the investigator to be a clinically significant change from Baseline or led to premature discontinuation of study treatment, dose modification, or other therapeutic intervention.
Time Frame: First dose to 30 days past last dose (Up to 36 Months)
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Alisertib (Phase 1 - Ovarian Cancer) | Alisertib (Phase 1 - Breast Cancer)
Number analyzed (Participants) | 38 | 11
participants
  Neutrophil count decreased | 3 | 0
  White blood cell count decreased | 1 | 1
  Aspartate aminotransferase increased | 3 | 1
  Alanine aminotransferase increased | 2 | 0
  Ammonia increased | 1 | 0
  Transaminases increased | 1 | 0
  Blood alkaline phosphatase increased | 1 | 1
  High density lipoprotein decreased | 1 | 0
  Urine output decreased | 1 | 0
  Granulocyte count decreased | 0 | 1

5. Primary Outcome: Phase 1: Number of Participants With Clinically Significant Vital Sign Findings
Description: Vital signs (blood pressure, pulse rate, and oral temperature) measurements were collected throughout the study.
Time Frame: First dose to 30 days past last dose (Up to 36 Months)
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Alisertib (Phase 1 - Ovarian Cancer) | Alisertib (Phase 1 - Breast Cancer)
Number analyzed (Participants) | 38 | 11
participants
  Pyrexia | 8 | 5
  Heart rate irregular | 1 | 0
  Blood pressure increased | 0 | 1
  Weight decreased | 3 | 0

6. Primary Outcome: Phase 1: Number of Participants With Hypersensitivity and Neurotoxicity
Time Frame: Baseline up to Month 36
Population: Explanation of how the number of participants for analysis was determined. Includes whether analysis was per protocol, intention to treat, or another method. Also provides relevant details such as imputation technique, as appropriate.
  Safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Alisertib (Phase 1 - Ovarian Cancer) | Alisertib (Phase 1 - Breast Cancer)
Number analyzed (Participants) | 38 | 11
participants
  Hypersensitivity | 1 | 0
  Neurotoxicity | 0 | 0

7. Primary Outcome: Phase 2: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date randomization for Phase 2 participants to the date of first documented progressive disease (PD) or death as assessed by the investigator using both RECIST 1.1 criteria and CA-125 criteria. PD is defined as 20% increase in the sum of the longest diameter of target lesions for measurable neoplastic disease or CA-125 criteria with elevated (>70 units/mL) levels on 2 occasions. CA 125 progression for participants with normal CA 125 levels is defined as a CA 125 level > 2 times the upper limit of normal and for participants with elevated values during the trial, is defined as a CA 125 level greater than 2 times the nadir value of CA 125.
Time Frame: At the end of Cycle 2 and at the completion of every 2 cycles until PD was documented or up to data cut-off: 12 August 2014 (approximately 24 months)
Population: The modified intent-to-treat (mITT) population was defined as all participants who were randomized and received at least 1 dose of any study drug. For a participant that has not progressed and has not died or has started the alternate therapy, PFS is censored at the last response assessment that is stable disease (SD) or better.
Measure: Median (80% Confidence Interval); unit: days
Groups:
- Paclitaxel 80 mg/m^2 (Phase 2): Paclitaxel 80 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 2.
Arm/Group | Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 (Phase 2) | Paclitaxel 80 mg/m^2 (Phase 2)
Number analyzed (Participants) | 73 | 69
days | 204 [175 to 230] | 142 [117 to 148]

8. Secondary Outcome: Phase 1: Combined Best Overall Response Rate (ORR) in Participants With Recurrent Ovarian Cancer or Breast Cancer
Description: Combined objective response rate is defined as the percentage of participants with Complete Response (CR) + Partial Response (PR) as assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1 or response by Cancer antigen (CA) 125 criteria. According to RECIST: CR is defined as disappearance of all target lesions and PR is defined as 30% decrease in the sum of the longest diameter of target lesions. CA 125 response criteria is defined as either: A 50% decrease from 2 initially elevated samples; the sample demonstrating the 50% decrease must have been confirmed by a fourth sample 28 days later (a total of 4 samples required) or A serial decrease of > 75% over 3 samples; the third sample was to be obtained 28 days after the second (a total of 3 samples required).
Time Frame: as for outcome 7
Population: Response evaluable population was defined as all participants who were randomized and had measurable disease according to RECIST or assessable disease by CA-125 criteria, who received at least 1 dose of any study drug, and who had at least 1 available post-Baseline response assessment as per either RECIST or CA-125 criteria.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Alisertib (Phase 1 - Ovarian Cancer) | Alisertib (Phase 1 - Breast Cancer)
Number analyzed (Participants) | 38 | 11
percentage of participants | 47 [36 to 59] | 55 [32 to 76]

9. Secondary Outcome: Cmax: Maximum Observed Concentration for Alisertib in Phase 1
Time Frame: Days 1 and 3 in Cycle 1: pre-dose and at multiple timepoints (up to 12 hours) post morning dose
Population: Pharmacokinetic (PK) analysis set for alisertib was defined as all participants in the phase 1 portion of the study for whom there was sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Alisertib 10 mg BID + Paclitaxel 80 mg/m^2: Alisertib (MLN8237) 10 mg, orally, twice daily (BID) on Days 1-3, 8-10 and 15-17, combined with weekly paclitaxel 80 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 1.
- Alisertib 20 mg BID + Paclitaxel 80 mg/m^2: Alisertib 20 mg, orally, twice daily (BID) on Days 1-3, 8-10 and 15-17, combined with weekly paclitaxel 80 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 1.
- Alisertib 20 mg BID + Paclitaxel 60 mg/m^2: Alisertib 20 mg, orally, twice daily (BID) on Days 1-3, 8-10 and 15-17, combined with weekly paclitaxel 60 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 1.
- Alisertib 30 mg BID + Paclitaxel 60 mg/m^2: Alisertib 30 mg, orally, twice daily (BID) on Days 1-3, 8-10 and 15-17, combined with weekly paclitaxel 60 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase
- Alisertib 40 mg BID + Paclitaxel 60 mg/m^2; Alisertib 50 mg BID + Paclitaxel 60 mg/m^2: Alisertib 10 mg, orally, twice daily (BID) on Days 1-3, 8-10 and 15-17, combined with weekly paclitaxel 80 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 1.
Arm/Group | Alisertib 10 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 30 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 50 mg BID + Paclitaxel 60 mg/m^2
Number analyzed (Participants) | 15 | 6 | 4 | 6 | 15 | 3
ng/mL
  Cycle1 (Day1) | 428.7 (189.59) | 766.8 (312.10) | 900.00 (392.17) | 1365.3 (466.51) | 1398.7 (607.70) | 1960.0 (515.65)
  Cycle1 (Day3) | 594.3 (228.46) | 1042.3 (280.95) | 871.3 (268.23) | 1708.5 (820.54) | 2493.4 (955.31) | 4456.7 (947.33)

10. Secondary Outcome: Tmax: Time to First Occurrence of Cmax for Alisertib in Phase 1
Time Frame: Days 1 and 3 in Cycle 1: pre-dose and at multiple timepoints (up to 12 hours) post morning dose
Population: PK analysis set for alisertib was defined as all participants in the phase 1 portion of the study for whom there was sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis.
Measure: Median (Full Range); unit: hour
Arm/Group | Alisertib 10 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 30 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 50 mg BID + Paclitaxel 60 mg/m^2
Number analyzed (Participants) | 15 | 6 | 4 | 6 | 15 | 3
hour
  Cycle 1, Day 1 | 3.0 (189.59) [1 to 5] | 3.1 (312.10) [2 to 4] | 2.6 (392.17) [2 to 3] | 2.5 (466.51) [2 to 9] | 3.0 (607.70) [2 to 9] | 2.0 (515.65) [2 to 9]
  Cycle 1, Day 3 | 2.2 (228.46) [0 to 5] | 3.0 (280.95) [1 to 3] | 3.5 (268.23) [2 to 5] | 2.0 (820.54) [1 to 4] | 2.0 (955.31) [1 to 9] | 2.0 (947.33) [2 to 3]

11. Secondary Outcome: AUC(Tau): Area Under the Concentration-Time Curve During a Dosing Interval for Alisertib in Phase 1
Time Frame: Days 1 and 3 in Cycle 1: pre-dose and at multiple timepoints (up to 12 hours) post morning dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL*hour(hr)
Arm/Group | Alisertib 10 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 30 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 50 mg BID + Paclitaxel 60 mg/m^2
Number analyzed (Participants) | 15 | 6 | 4 | 6 | 15 | 3
ng/mL*hour(hr)
  Cycle 1, Day 1 | 2519.3 (937.52) | 5175.0 (1766.11) | 5610.0 (2105.42) | 8581.7 (3225.64) | 9594.0 (4600.42) | 14666.7 (3707.20)
  Cycle 1, Day3 | 3966.7 (1112.11) | 7745.0 (2233.91) | 6155.0 (1737.69) | 12478.3 (6013.93) | 17557.3 (7856.30) | 35500.0 (12842.12)

12. Secondary Outcome: AUClast: Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Alisertib in Phase 1
Time Frame: Days 1 and 3 in Cycle 1: pre-dose and at multiple timepoints (up to 12 hours) post morning dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL*hr
Arm/Group | Alisertib 10 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 30 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 50 mg BID + Paclitaxel 60 mg/m^2
Number analyzed (Participants) | 15 | 6 | 4 | 6 | 15 | 3
ng/mL*hr
  Cycle 1, Day 1 | 2519.3 (937.52) | 5175.0 (1766.11) | 5610.0 (2105.42) | 8581.7 (3225.64) | 9594.0 (4600.42) | 14666.7 (3707.20)
  Cycle 1, Day 3 | 3966.7 (1112.11) | 7745.0 (2233.91) | 6155.0 (1737.69) | 12478.3 (6013.93) | 17557.3 (7856.30) | 35500.0 (12842.12)

13. Secondary Outcome: Cmax: Maximum Observed Concentration for Paclitaxel in Phase 1
Time Frame: Day 1 in Cycles 1 and 2: pre-infusion and at multiple timepoints (up to 47 hours) post-infusion
Population: PK analysis set for paclitaxel was defined as all participants in the phase 1 portion of the study for whom there was sufficient dosing and paclitaxel concentration time data to permit noncompartmental PK analysis. Number analyzed is the number of participants with evaluable data at the specified time-point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alisertib 10 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 30 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 50 mg BID + Paclitaxel 60 mg/m^2
Number analyzed (Participants) | 15 | 6 | 4 | 6 | 15 | 3
ng/mL
  Cycle 1, Day 1: number analyzed (Participants) | 15 | 6 | 4 | 5 | 15 | 3
  Cycle 1, Day 1 | 3097.3 (1114.51) | 3120.0 (447.75) | 2117.5 (745.54) | 2448.0 (988.65) | 1917.3 (528.32) | 1338.7 (617.94)
  Cycle 2, Day 1: number analyzed (Participants) | 13 | 6 | 3 | 6 | 13 | 2
  Cycle 2, Day 1 | 2654.6 (696.45) | 3231.7 (615.64) | 1733.3 (541.97) | 2478.3 (878.39) | 1492.7 (558.14) | 1750.0 (183.85)

14. Secondary Outcome: AUClast: Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Paclitaxel in Phase 1
Time Frame: Day 1 in Cycles 1 and 2: pre-infusion and at multiple timepoints (up to 47 hours) post-infusion
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL*hr
Arm/Group | Alisertib 10 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 30 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 50 mg BID + Paclitaxel 60 mg/m^2
Number analyzed (Participants) | 15 | 6 | 4 | 6 | 15 | 3
ng/mL*hr
  Cycle 1, Day 1: number analyzed (Participants) | 13 | 6 | 4 | 5 | 15 | 3
  Cycle 1, Day 1 | 4437.7 (1053.87) | 4825.0 (735.17) | 3355.0 (865.89) | 3366.0 (1139.25) | 2652.7 (651.32) | 2190.0 (387.43)
  Cycle 2, Day 1: number analyzed (Participants) | 12 | 6 | 3 | 5 | 13 | 2
  Cycle 2, Day 1 | 4061.7 (1298.86) | 5301.7 (1183.31) | 2660.0 (307.90) | 3056.0 (812.67) | 2231.5 (604.76) | 2460.0 (14.14)

15. Secondary Outcome: AUC∞: Area Under the Concentration-Time Curve From Time 0 to Infinity, Calculated Using the Observed Value of the Last Quantifiable Concentration for Paclitaxel in Phase 1
Time Frame: Day 1 in Cycles 1 and 2: pre-infusion and at multiple timepoints (up to 47 hours) post-infusion
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL*hr
Arm/Group | Alisertib 10 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 30 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 50 mg BID + Paclitaxel 60 mg/m^2
Number analyzed (Participants) | 15 | 6 | 4 | 6 | 15 | 3
ng/mL*hr
  Cycle 1, Day 1: number analyzed (Participants) | 9 | 5 | 3 | 4 | 11 | 2
  Cycle 1, Day 1 | 5317.8 (1052.40) | 5238.0 (812.26) | 3860.0 (824.20) | 3375.0 (1130.56) | 3175.5 (933.10) | 2535.0 (657.61)
  Cycle 2, Day 1: number analyzed (Participants) | 11 | 5 | 2 | 4 | 10 | 0
  Cycle 2, Day 1 | 4606.4 (1391.35) | 5584.0 (1367.51) | 3185.0 (176.78) | 3415.0 (1010.82) | 2680.0 (607.22) |

16. Secondary Outcome: t½: Terminal Half-Life for Paclitaxel in Phase 1
Time Frame: Day 1 in Cycles 1 and 2: pre-infusion and at multiple timepoints (up to 47 hours) post-infusion
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Alisertib 10 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 30 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 50 mg BID + Paclitaxel 60 mg/m^2
Number analyzed (Participants) | 15 | 6 | 4 | 6 | 15 | 3
hour
  Cycle 1, Day 1: number analyzed (Participants) | 11 | 5 | 3 | 5 | 11 | 2
  Cycle 1, Day 1 | 17.2 (4.20) | 17.5 (1.87) | 17.3 (4.16) | 13.9 (4.68) | 16.8 (6.83) | 18.4 (8.70)
  Cycle 2, Day 1: number analyzed (Participants) | 12 | 5 | 2 | 4 | 10 | 2
  Cycle 2, Day 1 | 17.0 (3.63) | 16.2 (5.05) | 17.3 (5.23) | 16.5 (4.32) | 13.3 (5.59) | 14.6 (2.19)

17. Secondary Outcome: CL: Total Clearance After Intravenous Administration, Calculated Using the Observed Value of the Last Quantifiable Concentration for Paclitaxel in Phase 1
Time Frame: Day 1 in Cycles 1 and 2: pre-infusion and at multiple timepoints (up to 47 hours) post-infusion
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Alisertib 10 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 30 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 50 mg BID + Paclitaxel 60 mg/m^2
Number analyzed (Participants) | 15 | 6 | 4 | 6 | 15 | 3
liter per hour
  Cycle 1, Day 1: number analyzed (Participants) | 9 | 5 | 3 | 4 | 11 | 2
  Cycle 1, Day 1 | 29.756 (6.8175) | 28.220 (5.1804) | 26.800 (7.5386) | 40.950 (17.5268) | 38.055 (13.7095) | 38.950 (11.2430)
  Cycle 2, Day 1: number analyzed (Participants) | 11 | 5 | 2 | 4 | 10 | 0
  Cycle 2, Day 1 | 35.827 (10.4005) | 28.240 (7.3748) | 33.900 (5.2326) | 34.250 (8.2614) | 42.440 (10.4296) |

18. Secondary Outcome: Vss: Volume of Distribution at Steady State for Paclitaxel in Phase 1
Time Frame: Day 1 in Cycles 1 and 2: pre-infusion and at multiple timepoints (up to 47 hours) post-infusion
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Alisertib 10 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 30 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 50 mg BID + Paclitaxel 60 mg/m^2
Number analyzed (Participants) | 15 | 6 | 4 | 6 | 15 | 3
liter
  Cycle 1, Day 1: number analyzed (Participants) | 9 | 5 | 3 | 4 | 11 | 2
  Cycle 1, Day 1 | 313.444 (118.6593) | 310.800 (86.9235) | 330.000 (208.8851) | 357.000 (158.1834) | 433.909 (179.7757) | 460.500 (103.9447)
  Cycle 2, Day 1: number analyzed (Participants) | 11 | 5 | 2 | 4 | 10 | 0
  Cycle 2, Day 1 | 391.364 (64.3137) | 283.200 (121.1123) | 413.500 (242.5376) | 377.000 (118.9650) | 372.600 (180.7332) |

19. Secondary Outcome: Vz: Volume of Distribution During the Terminal Disposition Phase for Paclitaxel in Phase 1
Time Frame: Day 1 in Cycles 1 and 2: pre-infusion and at multiple timepoints (up to 47 hours) post-infusion
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Alisertib 10 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 80 mg/m^2 | Alisertib 20 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 30 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 | Alisertib 50 mg BID + Paclitaxel 60 mg/m^2
Number analyzed (Participants) | 15 | 6 | 4 | 6 | 15 | 3
liter
  Cycle 1, Day 1: number analyzed (Participants) | 9 | 5 | 3 | 4 | 11 | 2
  Cycle 1, Day 1 | 705.000 (179.0223) | 721.600 (203.8021) | 694.000 (352.1534) | 850.500 (291.0401) | 872.727 (328.6202) | 956.500 (188.7975)
  Cycle 2, Day 1: number analyzed (Participants) | 11 | 5 | 2 | 4 | 10 | 0
  Cycle 2, Day 1 | 829.364 (156.6060) | 663.200 (321.3070) | 865.500 (388.2016) | 777.250 (103.7027) | 733.000 (208.4898) |

20. Secondary Outcome: Phase 2: Combined Best Overall Response Rate (ORR)
Description: as for outcome 8
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 (Phase 2) | Paclitaxel 80 mg/m^2 (Phase 2)
Number analyzed (Participants) | 67 | 64
percentage of participants | 60 [51 to 68] | 52 [43 to 60]

21. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documentation of a response to the date of first documentation of PD or the last response assessment that is stable disease (SD) or better for a participant who started alternate therapy without progression. PD is defined as 20% increase in the sum of the longest diameter of target lesions for measurable neoplastic disease or per CA-125 criteria with elevated (>70 units/mL) levels on 2 occasions. CA 125 progression for participants with normal CA 125 levels is defined as a CA 125 level > 2 times the upper limit of normal and for participants with elevated values during the trial, is defined as a CA 125 level greater than 2 times the nadir value of CA 125. A responder that did not experience disease progression is censored at the last response assessment that is SD.
Time Frame: Up to data-cut off: 12 August 2014 (approximately 24 months)
Population: Participants from Response evaluable population, all participants who were randomized and had measurable disease according to RECIST 1.1 or assessable disease by CA-125 criteria, who received at least 1 dose of any study drug, and who had at least 1 available post-Baseline response assessment per RECIST 1.1 or CA-125 criteria, who were responders.
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 (Phase 2) | Paclitaxel 80 mg/m^2 (Phase 2)
Number analyzed (Participants) | 40 | 33
days | 201 [181 to 218] | 169 [120 to 231]

22. Secondary Outcome: Phase 2: Time to Disease Progression (TTP)
Description: TTP was defined as the time from the date of randomization to the date of first documentation of PD. PD is defined as 20% increase in the sum of the longest diameter of target lesions for measurable neoplastic disease or per CA-125 criteria with elevated (>70 units/mL) levels on 2 occasions. CA 125 progression for participants with normal CA 125 levels is defined as a CA 125 level > 2 times the upper limit of normal and for participants with elevated values during the trial, is defined as a CA 125 level greater than 2 times the nadir value of CA 125.
Time Frame: Up to data-cut off: 12 August 2014 (approximately 24 months)
Population: mITT Population was defined as all participants who were randomized and received at least 1 dose of any study drug. For a participant that has not progressed, TTP is censored at the last response assessment that is SD or better
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 (Phase 2) | Paclitaxel 80 mg/m^2 (Phase 2)
Number analyzed (Participants) | 73 | 69
days | 204 [175 to 232] | 142 [117 to 161]

23. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time form the date of the randomization to the date of death.
Time Frame: Up to data-cut off: 12 August 2014 (approximately 24 months)
Population: mITT Population was defined as all participants who were randomized and received at least 1 dose of any study drug. For a participant that is alive, OS will be censored at the last known date.
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 (Phase 2) | Paclitaxel 80 mg/m^2 (Phase 2)
Number analyzed (Participants) | 73 | 69
days | NA [NA to NA] — Median, upper and lower limits of CI were not reached due to low number of participants with events. | NA [NA to NA] — Median, upper and lower limits of CI were not reached due to low number of participants with events.

24. Secondary Outcome: Phase 2: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: as for outcome 3
Time Frame: First dose to 30 days past last dose (Up to 27 Months)
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 (Phase 2) | Paclitaxel 80 mg/m^2 (Phase 2)
Number analyzed (Participants) | 73 | 69
participants
  AEs | 73 | 66
  SAEs | 30 | 19

25. Secondary Outcome: Phase 2: Number of Participants With Clinically Significant Laboratory Values
Description: as for outcome 4
Time Frame: First dose to 30 days past last dose (Up to 27 Months)
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Groups:
- Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 (Phase 2): Alisertib 40 mg, orally, BID on Days 1-3, 8-10 and 15-17, combined with weekly paclitaxel 60 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 2 (Up to 28 cycles).
Arm/Group | Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 (Phase 2) | Paclitaxel 80 mg/m^2 (Phase 2)
Number analyzed (Participants) | 73 | 69
participants
  Neutrophil count decreased | 14 | 4
  White blood cell count decreased | 6 | 1
  Lymphocyte count decreased | 1 | 1
  Aspartate aminotransferase increased | 1 | 3
  Alanine aminotransferase increased | 1 | 4
  Gamma-glutamyltransferase increased | 0 | 1
  Blood alkaline phosphatase increased | 2 | 2
  Haemoglobin decreased | 3 | 1
  Blood magnesium decreased | 0 | 3
  Blood creatinine increased | 1 | 2
  Platelet count decreased | 2 | 0
  International normalised ratio increased | 1 | 0
  Blood albumin decreased | 1 | 0
  Troponin T increased | 0 | 1

26. Secondary Outcome: Phase 2: Number of Participants With Clinically Significant Vital Sign Findings
Description: Vital signs (blood pressure, pulse rate, and oral temperature) measurements were collected throughout the study.
Time Frame: First dose to 30 days past last dose (Up to 27 Months)
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Alisertib 40 mg BID + Paclitaxel 60 mg/m^2 (Phase 2) | Paclitaxel 80 mg/m^2 (Phase 2)
Number analyzed (Participants) | 73 | 69
participants
  Pyrexia | 15 | 8
  Heart rate increased | 1 | 0
  Blood pressure increased | 1 | 0
  Weight decreased | 8 | 2

27. Other Pre Specified Outcome: Banked Tumor Specimens for Candidate Markers of Response to Alisertib and Taxanes
Time Frame: Up to 24 Months
Population: This Outcome Measure was originally registered as a Secondary but this Outcome Measure was Exploratory and no data was collected.
Arm/Group | Alisertib + Paclitaxel (Phase 1)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Phase 1: First dose to 30 days past last dose (Up to 36 Months); Phase 2: First dose to 30 days past last dose (Up to 27 Months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Alisertib (Phase 1 - Ovarian Cancer): Alisertib (MLN8237) 10 mg, orally, twice daily (BID) on Days 1-3, 8-10 and 15-17, combined with weekly paclitaxel 80 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 1.
- Alisertib (Phase 1 - Breast Cancer): Alisertib 20 mg, orally, twice daily (BID) on Days 1-3, 8-10 and 15-17, combined with weekly paclitaxel 80 mg/m^2, intravenous infusion, weekly (Days 1, 8, 15) in 28-day cycles in Phase 1.
Arm/Group | Alisertib (Phase 1 - Ovarian Cancer) | Alisertib (Phase 1 - Breast Cancer) | Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 (Phase 2) | Paclitaxel 80 mg/m^2 (Phase 2)
Serious Adverse Events (participants affected / at risk) | 13/38 | 2/11 | 30/73 | 19/69
Other Adverse Events (participants affected / at risk) | 38/38 | 11/11 | 73/73 | 64/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alisertib (Phase 1 - Ovarian Cancer) (N=38) | Alisertib (Phase 1 - Breast Cancer) (N=11) | Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 (Phase 2) (N=73) | Paclitaxel 80 mg/m^2 (Phase 2) (N=69)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (9) | 0 (0) | 9 (9) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (7) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (4) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (4) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) — One treatment-emergent death occurred during treatment with alisertib and paclitaxel and was not related.
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abscess soft tissue (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) — One treatment-emergent death occurred during treatment with paclitaxel and was not related.
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postrenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraneoplastic dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alisertib (Phase 1 - Ovarian Cancer) (N=38) | Alisertib (Phase 1 - Breast Cancer) (N=11) | Alisertib 40 mg BID+ Paclitaxel 60 mg/m^2 (Phase 2) (N=73) | Paclitaxel 80 mg/m^2 (Phase 2) (N=69)
Diarrhoea (Gastrointestinal disorders) | 27 (49) | 8 (11) | 46 (96) | 15 (19)
Nausea (Gastrointestinal disorders) | 23 (33) | 5 (6) | 32 (54) | 32 (46)
Stomatitis (Gastrointestinal disorders) | 15 (32) | 8 (10) | 46 (91) | 6 (8)
Constipation (Gastrointestinal disorders) | 15 (22) | 3 (4) | 26 (33) | 17 (23)
Abdominal pain (Gastrointestinal disorders) | 12 (19) | 3 (3) | 21 (39) | 20 (26)
Vomiting (Gastrointestinal disorders) | 13 (42) | 4 (4) | 20 (31) | 18 (25)
Abdominal pain upper (Gastrointestinal disorders) | 3 (5) | 1 (1) | 11 (12) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 1 (1) | 9 (12) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2) | 9 (10) | 4 (4)
Ascites (Gastrointestinal disorders) | 3 (3) | 1 (1) | 8 (11) | 5 (7)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 0 (0) | 9 (10) | 2 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 0 (0) | 6 (7) | 4 (5)
Oral pain (Gastrointestinal disorders) | 5 (6) | 0 (0) | 6 (6) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 5 (6) | 2 (2) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 6 (9) | 1 (3) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (9) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (6) | 1 (2)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (4)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Fatigue (General disorders) | 26 (29) | 8 (10) | 43 (82) | 31 (37)
Oedema peripheral (General disorders) | 15 (24) | 3 (3) | 12 (15) | 18 (25)
Pyrexia (General disorders) | 8 (11) | 4 (7) | 13 (18) | 7 (10)
Asthenia (General disorders) | 5 (6) | 2 (2) | 10 (20) | 8 (11)
Chills (General disorders) | 10 (12) | 0 (0) | 6 (6) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2) | 3 (4) | 0 (0)
Catheter site pain (General disorders) | 3 (5) | 0 (0) | 2 (2) | 1 (1)
Peripheral swelling (General disorders) | 2 (3) | 0 (0) | 2 (4) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 24 (100) | 10 (58) | 52 (179) | 10 (17)
Anaemia (Blood and lymphatic system disorders) | 22 (37) | 7 (13) | 33 (61) | 20 (36)
Leukopenia (Blood and lymphatic system disorders) | 20 (47) | 8 (32) | 11 (27) | 3 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (17) | 4 (7) | 1 (2)
Granulocytopenia (Blood and lymphatic system disorders) | 3 (4) | 1 (4) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (29) | 5 (6) | 28 (36) | 22 (24)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 2 (2) | 5 (5) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 5 (5) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 5 (5) | 2 (4)
Erythema (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1) | 2 (2) | 2 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
Skin lesion (Skin and subcutaneous tissue disorders) | 6 (12) | 0 (0) | 1 (3) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (4) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (10) | 0 (0) | 0 (0) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 8 (8) | 4 (4) | 12 (15) | 13 (16)
Headache (Nervous system disorders) | 6 (9) | 1 (1) | 8 (11) | 13 (22)
Dizziness (Nervous system disorders) | 8 (14) | 0 (0) | 10 (16) | 6 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 2 (2) | 9 (9) | 8 (9)
Dysgeusia (Nervous system disorders) | 7 (9) | 0 (0) | 4 (4) | 5 (6)
Somnolence (Nervous system disorders) | 2 (3) | 1 (1) | 7 (9) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 5 (8)
Restless legs syndrome (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3) | 2 (2)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 3 (3) | 17 (20) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 3 (3) | 9 (10) | 11 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 1 (1) | 6 (6) | 7 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 1 (1) | 6 (7) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 3 (5) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 4 (5) | 2 (2) | 1 (1) | 1 (1)
Lacrimation increased (Eye disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Visual impairment (Eye disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Eye pruritus (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 2 (4) | 0 (0) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meibomian gland dysfunction (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (15) | 2 (7) | 9 (11) | 9 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (18) | 3 (3) | 7 (9) | 6 (9)
Fall (Injury, poisoning and procedural complications) | 8 (14) | 0 (0) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (14) | 1 (1) | 8 (9) | 5 (6)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (7) | 0 (0) | 4 (4) | 7 (9)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (10) | 1 (1) | 4 (4) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (5) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 4 (5) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (9) | 0 (0) | 0 (0) | 1 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (4) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 (8) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 5 (5) | 1 (1) | 1 (1) | 2 (2)
Palpitations (Cardiac disorders) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 (4) | 0 (0) | 0 (0) | 2 (2)
Genital discomfort (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 12 (17) | 2 (2) | 15 (18) | 8 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (8) | 4 (5) | 13 (27) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (16) | 3 (3) | 8 (9) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 7 (8) | 0 (0) | 8 (9) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (3) | 2 (2) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 3 (3) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 3 (4) | 0 (0) | 3 (3) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Seasonal allergy (Immune system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 1 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (3) | 5 (5)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 4 (12) | 3 (9)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 1 (1) | 3 (5) | 1 (2)
Hot flush (Vascular disorders) | 3 (4) | 0 (0) | 1 (1) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 4 (5) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 2 (2) | 8 (8) | 7 (8)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1) | 11 (11) | 7 (9)
Depression (Psychiatric disorders) | 4 (4) | 1 (1) | 6 (7) | 4 (4)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (4) | 0 (0) | 13 (22) | 4 (5)
Weight decreased (Investigations) | 3 (3) | 0 (0) | 8 (11) | 2 (2)
White blood cell count decreased (Investigations) | 1 (2) | 1 (6) | 6 (14) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (2) | 1 (2) | 3 (4)
Alanine aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 1 (2) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (2) | 2 (3) | 2 (3)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Granulocyte count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 11 (29) | 4 (8) | 11 (20) | 4 (7)
Upper respiratory tract infection (Infections and infestations) | 11 (24) | 4 (4) | 3 (4) | 4 (5)
Sinusitis (Infections and infestations) | 3 (10) | 3 (3) | 1 (1) | 2 (2)
Oral candidiasis (Infections and infestations) | 4 (4) | 0 (0) | 2 (2) | 1 (1)
Oral herpes (Infections and infestations) | 2 (4) | 0 (0) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Folliculitis (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Cellulitis (Infections and infestations) | 2 (5) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Localised infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.